CLINICAL TRIAL: NCT00277498
Title: A 12-Week, Randomized, Double-Masked, Parallel Group Comparison Of Xalacom Given In The Evening, Xalatan Given In The Evening, And Timolol Given In The Morning In Patients With Open Angle Glaucoma Or Ocular Hypertension In The United States.
Brief Title: A 12-week, Randomized, Double-masked, Parallel Group Comparison of Evening Dosing With Xalacom in Subjects With Glaucoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A6641044
Record Dates: First submitted 2006-01-13; First posted 2006-01-16 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2008-06

CONDITIONS: Open Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Xalacom; Latanoprost; Timolol

INTERVENTIONS:
Drug: Xalacom
Drug: Xalatan
Drug: Timolol

SUMMARY:
To demonstrate statistical superiority of the combination of latanoprost and timolol to the individual therapy of latanoprost and timolol based on intraocular pressure measurements at 8 AM, 10 AM, 4 PM at weeks 2, 6 and 12.

ELIGIBILITY:
Inclusion Criteria:

* Uni- or bilateral diagnosis of primary open angle glaucoma or ocular hypertension on beta-blocker monotherapy or dual therapy in which at least one medication is a beta-blocker for at least 4 weeks prior to screening

Exclusion Criteria:

* Closed/ barely open anterior chamber angle or history of acute angle closure glaucoma.
* History of ALT (Argon Laser Trabeculoplasty) or SLT(selective Laser) within 3 months prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 528
Dates: Start 2005-12; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
The mean IOP measurements obtained in the study eye at each time point.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (55):
- United States (55):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Flagstaff, Arizona
  - Pfizer Investigational Site, Artesia, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Newport Beach, California
  - Pfizer Investigational Site, Sacramento, California
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, Colorado Springs, Colorado
  - Pfizer Investigational Site, Gainesville, Florida
  - Pfizer Investigational Site, Lecanto, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Panama City, Florida
  - Pfizer Investigational Site, Idaho Falls, Idaho
  - Pfizer Investigational Site, Bourbonnais, Illinois
  - Pfizer Investigational Site, Calumet City, Illinois
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Evansville, Indiana
  - Pfizer Investigational Site, Madison, Indiana
  - Pfizer Investigational Site, New Albany, Indiana
  - Pfizer Investigational Site, Newburgh, Indiana
  - Pfizer Investigational Site, Iowa City, Iowa
  - Pfizer Investigational Site, Wichita, Kansas
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Bangor, Maine
  - Pfizer Investigational Site, Reading, Massachusetts
  - Pfizer Investigational Site, Ann Arbor, Michigan
  - Pfizer Investigational Site, Detroit, Michigan
  - Pfizer Investigational Site, Stillwater, Minnesota
  - Pfizer Investigational Site, Creve Coeur, Missouri
  - Pfizer Investigational Site, Kansas City, Missouri
  - Pfizer Investigational Site, Warrensburg, Missouri
  - Pfizer Investigational Site, Washington, Missouri
  - Pfizer Investigational Site, Piscataway, New Jersey
  - Pfizer Investigational Site, Princeton, New Jersey
  - Pfizer Investigational Site, Brooklyn, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Durham, North Carolina
  - Pfizer Investigational Site, Greensboro, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Roseburg, Oregon
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Reading, Pennsylvania
  - Pfizer Investigational Site, Wyomissing, Pennsylvania
  - Pfizer Investigational Site, Charleston, South Carolina
  - Pfizer Investigational Site, Maryville, Tennessee
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, El Paso, Texas
  - Pfizer Investigational Site, Fort Worth, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Fredericksburg, Virginia
  - Pfizer Investigational Site, Seattle, Washington

REFERENCES:
- [Derived] Higginbotham EJ, Olander KW, Kim EE, Grunden JW, Kwok KK, Tressler CS; United States Fixed-Combination Study Group. Fixed combination of latanoprost and timolol vs individual components for primary open-angle glaucoma or ocular hypertension: a randomized, double-masked study. Arch Ophthalmol. 2010 Feb;128(2):165-72. doi: 10.1001/archophthalmol.2009.384. PMID 20142538
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6641044&StudyName=A%2012-week%2C%20randomized%2C%20double-masked%2C%20parallel%20group%20comparison%20of%20evening%20dosing%20with%20Xalacom%20in%20subjects%20with%20glaucoma